CLINICAL TRIAL: NCT04940494
Title: Incidence and Risk Factors for Anal Incontinence After Obstetrical Anal Sphincter Injury
Brief Title: Anal Incontinence After Obstetrical Anal Sphincter Injury
Acronym: INCONT-LOSA
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-A01128-33
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Obstetric Trauma; Anal Sphincter Injury; Anal Incontinence
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: collection of data — collection of data for all Obstetrical Anal Sphincter Injury women (score of quality of life, experimenting anal incontinence...)

SUMMARY:
Obstetrical Anal Sphincter Injury is an identified risk factor for anal incontinence. The mechanisms and the risk factors for anal incontinence in Obstetrical Anal Sphincter Injury women are not well known.

Anal incontinence in such women is not well documented and probably underestimated. Cohort studies estimated that up to 53% of Obstetrical Anal Sphincter Injury women are incontinent but that most of them does not complain their doctor.

ELIGIBILITY:
Inclusion Criteria:

* Childbirth between 2005 January 1st and 2019 December 31th
* Obstetrical Anal Sphincter Injury -≥ 18 y

Exclusion Criteria:

* Patients' refusal
* lost of view or deceased
* anal incontinence before the Obstetrical Anal Sphincter Injury

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women that gave birth between 2005 January 1st and 2019 December 31th and that accept to respond to the survey
Sampling Method: Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
anal incontinence | from the childbirth to the day of survey (2 to 16 years after childbirth)
  loss of stool or gas ≥1/week during ≥1 month

SECONDARY OUTCOMES:
Incidence of anal incontinence | Incidence of anal incontinence the date of the survey (2 to 16 years after childbirth)
  AI graded by the St Mark Score
cinetic of AI occurence | from the childbirth to the date of the survey (2 to 16 years after childbirth)
  all the resolutive episodes of occurence of anal incontinence are reported
Quality of life with fecal incontinence quality of life score | the date of the survey (2 to 16 years after childbirth)
  fecal incontinence quality of life score
Expectation of the women in term of information | the date of the survey (2 to 16 years after childbirth)
  2 questions on the expectation of the women in term of information towards the Obstetrical Anal Sphincter Injury

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien VENARA, M.D., Principal Investigator — University Hospital of Angers
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rebmann E, Hamel JF, Helbert C, Lemasson F, Legendre G, Venara A. Anal incontinence after obstetrical anal sphincter injury significantly impacts quality of life for women: a cohort study. Langenbecks Arch Surg. 2024 Feb 17;409(1):67. doi: 10.1007/s00423-024-03257-4. PMID 38368278